CLINICAL TRIAL: NCT04486755
Title: A Phase I Dose Escalation Study of Hypofractionated Accelerated Pelvic Nodal Radiotherapy Delivered With A Simultaneously Integrated Prostate Boost For Patients With Localized, Intermediate- And High-Risk Prostate Cancer (GCC 2048)
Brief Title: Hypofractionated Accelerated Pelvic Nodal Radiotherapy (GCC 2048)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HP-00091499
Record Dates: First submitted 2020-07-15; First posted 2020-07-27 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma
Keywords: Prostate; Hypofractionated Radiation Therapy; Prostate Cancer; Radiotherapy; Proton Therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: A modified 3+3 study design will be employed to determine the dose-fractionation schedule that results in less than 33% dose limiting toxicity. One de-escalation will be allowed if the initial dose-fractionation schedule results in too high a frequency of dose limiting toxicities. A total of 6 patients will be treated following the dose-fractionation schedule that is recommended for further study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Level 1 (Experimental): Dose schedules were calculated to maintain similar BED for late normal tissue injury (α/β= 3.0 Gy), with an increased BED for PC (α/β= 1.5Gy). Patients be treated with 20 fractions. A total of 6 patients will be treated at the dose that is determined to be Maximum Tolerated Dose.
  Interventions: Radiation: Hypofractionated Radiation Therapy
- Dose Level 2 (Experimental): Dose schedules were calculated to maintain similar BED for late normal tissue injury (α/β= 3.0 Gy), with an increased BED for PC (α/β= 1.5Gy). Patients be treated with 16 fractions. A total of 6 patients will be treated at the dose that is determined to be Maximum Tolerated Dose.
  Interventions: Radiation: Hypofractionated Radiation Therapy
- Dose Level 3 (Experimental): Dose schedules were calculated to maintain similar BED for late normal tissue injury (α/β= 3.0 Gy), with an increased BED for PC (α/β= 1.5Gy). Patients be treated with 12 fractions. A total of 6 patients will be treated at the dose that is determined to be Maximum Tolerated Dose.
  Interventions: Radiation: Hypofractionated Radiation Therapy

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — All patients RT will be delivered utilizing pencil beam scanning proton therapy. Radiation treatment will be delivered 4 days per week.

SUMMARY:
A phase I trial to determine the safety of delivering three sequentially shorter RT schedules (20, 16, and 12 fractions) of HypoFx pelvic nodal RT in combination with a HypoFx, simultaneous integrated boost (SIB) to the prostate that have been designed to incrementally increased the biological equivalent dose (BED) to prostate cancer, while maintaining a constant BED to normal tissue toxicity.

DETAILED DESCRIPTION:
Outcomes for patients with unfavorable intermediate-risk and high-risk prostate cancer (PC) have been historically poor and are now known to require multimodality treatment. A standard non-surgical treatment option for patients with localized, intermediate and high-risk PC is radiation therapy (RT) in combination with short- or long-term androgen deprivation therapy (ADT).

The benefit of pelvic nodal RT in this setting is unclear, previous studies have been equivocal. There is a growing body of evidence to demonstrate that use of hypofractionated (HypoFx) RT may be a safe method for increasing the dose of RT, while also decreasing normal tissue toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age is ≥ 18 years
2. Pathologically (histologically or cytologically) proven diagnosis of prostatic adenocarcinoma within 180 days of registration.
3. Patient's with intermediate to high risk prostate cancer and must be recommended to undergo pelvic as well as prostatic irradiation.
4. History/physical examination (to include at a minimum digital rectal examination of the prostate and examination of the skeletal system and abdomen) within 90 days prior to registration.
5. Clinically negative lymph nodes as established by imaging (pelvic ± abdominal CT or MR), (but not by nodal sampling, or dissection) within 120 days prior to registration.

   • Patients with lymph nodes equivocal or questionable by imaging are eligible if the nodes are ≤ 1.5 cm.
6. No evidence of bone metastases (M0) on bone scan within 120 days prior to registration.

   • Equivocal bone scan findings are allowed if plain films (or CT or MRI) are negative for metastasis.
7. Baseline serum PSA value performed within 12 weeks (90 days) prior to registration.
8. ECOG Performance Status 0-1
9. Patient must be able to provide study specific informed consent prior to study entry.

Exclusion Criteria:

1. Evidence of distant metastases
2. Regional lymph node involvement
3. Previous radical surgery (prostatectomy), cryosurgery, or HIFU (High-intensity focused ultrasound) for prostate cancer
4. Previous pelvic irradiation or prostate brachytherapy
5. Planned prostate brachytherapy boost
6. Previous or concurrent cytotoxic chemotherapy for prostate cancer
7. Severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.
8. Patients are excluded if they have a history of autoimmune disease that, in the opinion of the treating physician would be a contraindication to pelvic radiation (e.g., active systemic lupus, progressive scleroderma)
9. Patients receiving full-dose anticoagulation or clopidogrel

   • Patients taking 81 mg Aspirin po daily may are still eligible for the study
10. Patients with a history of prior small bowel ulceration

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-11-19 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
HypoFx RT schedule that results in <33% acute dose-limiting toxicity with accelerated, HypoFx pelvic nodal RT | Within 90 days of completing RT
  The frequency of all observed acute GI, GU, hematologic, and neurologic dose limiting toxicities by CTCAE v5 grade will be tabulated. DLT is defined as treatment-related: Grade ≥3 GI (small bowel or rectal) toxicity, Grade ≥3 GU toxicity, Grade ≥3 hematologic, Grade ≥3 neurologic toxicity, or any grade 5 treatment-related adverse events.

SECONDARY OUTCOMES:
Frequency of acute and late GI, GU, hematologic, and neurologic toxicity for each dose cohort | Acute (within 90 days completing RT), Late (occurring > 90 days from treatment), 3-months, 6 months, 1-year and 2 years
  The frequency of the maximum grade acute (within 90 days completing RT) and late (occurring > 90 days from treatment) GI (small bowel and rectal), GU, hematologic, and neurologic toxicities at 3-months, 6 months, 1-year and 2 years for each dose cohort using National Cancer Institute Common Terminology Criteria v.5.0 (NCI CTCAE v5).
Dose volume histogram (DVH) parameters | Within 90 days of completing RT
  A dose-volume histogram is a histogram relating radiation dose to tissue volume in radiation therapy planning.
Evaluate the duration of biochemical progression-free survival | 2 years after completing RT
  The duration of bPFS will be measured from the end of RT until either PSA recurrence or death due to any cause and summarized for the expanded cohort of patients treated at the maximum total dose (MTD). PSA recurrence is defined by the Phoenix definition of biochemical failure (PSA nadir + 2 ng/mL).
Patient Reported Outcomes (PROs) related to urinary and bowel function | 1 month after completion of treatment, every 3 months for year 1, and every 6 months during Year 2
  Quality of life will be assessed with the validated Expanded Prostate Cancer Index Composite (EPIC) questionnaire.
Patient Reported Outcomes (PROs) related to urinary function | 1 month after completion of treatment, every 3 months for year 1, and every 6 months during Year 2
  The International Prostate System Score (IPSS) questionnaire will be used for urinary function.
Patient Reported Outcomes (PROs) related to urinary and bowel function | 1 month after completion of treatment, every 3 months for year 1, and every 6 months during Year 2
  The PRO-CTCAE questionnaire measures patient-reported bowel, urinary and sexual function.

CONTACTS AND LOCATIONS:
Locations (1):
- Maryland Proton Treatment Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No